CLINICAL TRIAL: NCT00941655
Title: Prospective Randomized Trial Comparing Gastrectomy, Metastasectomy Plus Systemic Therapy Versus Systemic Therapy Alone: GYMSSA Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Udo Rudloff, M.D., Principal investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090189; 09-C-0189
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Gastric Cancer
Keywords: Gastric Carcinoma; Chemotherapy; Liver Tumors; Peritoneal Tumors; Metastatic Gastric Cancer; Stomach Cancer; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Surgery + HIPEC + Systemic Chemotherapy (Experimental): Surgery -gastric resection, metastasectomy, and heated intraperitoneal chemotherapy with Fluouracil (5-FU) 400 mg/m^2 intravenous (IV) over 5 minutes. Leucovorin 20 mg/m^2 IV and Oxaliplatin 460 mg/m^2 diluted in 2.0 L/m^2 of dextrose 5% in water (D5W) given as a heated intraperitoneal perfusion.
  Systemic chemotherapy - Irinotecan 165 mg/m^2 IV over 90 minutes, Oxaliplatin 85 mg/m^2 over 120 minutes, Leucovorin 200 mg/m^2 IV 120 minutes, 5FU 3200 mg/m^2 continuous IV infusion over 48 hours.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: 5-Fluorouracil; Drug: Leucovorin; Procedure: Gastrectomy and/or metastasectomy
- Systemic Chemotherapy Alone (Experimental): Irinotecan 165 mg/m^2 IV over 90 minutes, Oxaliplatin 85 mg/m^2 over 120 minutes, Leucovorin 200 mg/m^2 IV 120 minutes, 5FU 3200 mg/m^2 continuous IV infusion over 48 hours.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: 5-Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 460 mg/m^2 diluted in 2.0 L/m^2 of dextrose 5% in water (D5W) given as a heated intraperitoneal perfusion.
  Systemic chemotherapy - Oxaliplatin 85 mg/m^2 over 120 minutes,
  Other Names: Eloxatin
Drug: Irinotecan — Irinotecan 165 mg/m^2 IV over 90 minutes
  Other Names: Camptosar
Drug: 5-Fluorouracil — Surgery and heated intraperitoneal chemotherapy with Fluouracil (5-FU) 400 mg/m^2 intravenous (IV) over 5 minutes.
  systemic chemotherapy -3200 mg/m^2 continuous intravenous over 48 hours.
  Other Names: Efudex; Adracil; Carac
Drug: Leucovorin — surgery and heated intraperitoneal chemotherapy -20 mg/m^2 intravenous over 5 minutes.
  systemic chemotherapy - 200 mg/m^2 intravenous over 120 minutes.
  Other Names: Folinic acid
Procedure: Gastrectomy and/or metastasectomy — Gastrectomy: tumor resection and a bypass; palliative treatment for pain, bleeding, obstruction and/or if deemed in the best interest of the patient.
  Metastasectomy: anatomical segmental resection to render the patient no evidence of disease (NED) with at least 1cm negative margins when possible, followed by systemic chemotherapy.
  Arms: Surgery + HIPEC + Systemic Chemotherapy

SUMMARY:
Background:

* Gastric (stomach) cancer is a rare cancer. In most cases, by the time it has been diagnosed it has spread to other organs in the body and the chance of a cure is very small. The standard treatment for gastric cancer is a combination of chemotherapy drugs.
* Researchers are interested in finding out if surgically removing all tumors before beginning chemotherapy for stomach cancer can slow or halt its spread better than giving chemotherapy alone.

Objectives:

- To determine whether tumor removal surgery followed by chemotherapy is more effective in treating gastric cancer than chemotherapy given alone.

Eligibility:

- Patients 18 years of age and older who have been diagnosed with gastric cancer.

Design:

* All patients will undergo an initial physical examination, blood tests, imaging scans, and a laparoscopy to determine the extent of the disease.
* Half of the participants will be assigned to have surgery first and then chemotherapy; the other half will be assigned to have chemotherapy alone.

  * The surgery-plus-chemotherapy group will have major surgery to remove all tumors in the stomach and abdominal area, followed by a recovery time of up to 4 weeks. Chemotherapy will begin 6 to 8 weeks after surgery.
  * The chemotherapy-only group will begin treatment within 2 weeks of laparoscopy.
* All patients will receive four chemotherapy drugs: 5-Fluorouracil, leucovorin, oxaliplatin, and irinotecan. The drugs are given intravenously over 2 days every 2 weeks (one cycle) for 12 cycles (about 6 months), either at the National Institutes of Health (NIH) Clinical Center or at home with a referring oncologist. Patients in the surgery group who have tumors in the peritoneum will receive an additional set of chemotherapy drugs in a separate treatment.
* During the chemotherapy cycles, patients will provide blood samples approximately once a week and will have physical examinations and scans on a regular basis.
* Patients will return to the NIH Clinical Center for follow-up visits about every 4 months for 2 years, then every 6 months for 3 years and yearly thereafter.

DETAILED DESCRIPTION:
Background:

* The standard of care for metastatic gastric cancer (MGC) is systemic therapy resulting in median survival of 6-12 months and rare survivors of up to three years.
* For patients with limited MGC, retrospective studies have shown improved overall survival following gastrectomy and/or metastasectomy plus systemic therapy (e.g. median survival after liver resection for metastatic gastric cancer of 15-37 months, with a five year survival rate of 25%).
* This prospective randomized trial for patients with MGC and limited metastases is designed to compare two therapeutic approaches-gastrectomy with metastasectomy plus systemic therapy (GYMS) vs. systemic therapy alone (SA)-- and to evaluate outcome in light of selection criteria to define those patients who may benefit from the more aggressive approach.

Objectives:

Primary Objective:

- To compare two therapeutic approaches--GYMS vs. SA--in terms of overall survival in patients with limited MGC.

Secondary Objectives:

* To analyze selection criteria for patients who might benefit from the GYMS approach.
* To determine progression-free survival in both arms.

Eligibility:

* MGC with limited metastatic disease thought to be resectable to no evidence of disease.
* 18 years old or greater with an Eastern Cooperative Oncology Group (ECOG) 0-2
* Laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to surgery

Design:

* Patients will be randomized to receive gastrectomy and metastasectomy followed by systemic chemotherapy (GYMS) or systemic chemotherapy (SA) alone and will be stratified based on sites of metastatic disease, previous therapy and disease free interval.
* Patients in both arms will receive the FOLFOXIRI regimen (5-FU, leucovorin, oxaliplatin and irinotecan)
* No cross over will be allowed.
* Survival analysis will be done in intention to treat fashion from time of randomization.
* Based on estimated 12 and 20 months overall survival for the SA and the GYMS arms respectively, 68 patients per arm (power=0.80, 0.05 two-tailed log-rank test) will be enrolled. Patients will be recruited over 6 years and followed for an additional 2 years from the date of entry of the last patient.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Histologically or cytologically confirmed gastric adenocarcinoma.
2. Metastatic disease must be measurable by computed tomography (CT) and/or magnetic resonance imaging (MRI)

   Or

   There must be a history of positive peritoneal washings or carcinomatosis
3. All disease should be deemed resectable to negative margins (NED) based on imaging studies.

   Note: Patients with both pulmonary and peritoneal metastases will be enrolled at the discretion of the Principal Investigator.
   * Esophageal invasion < 4cm that does not require thoracotomy (Seiwert II and III lesions).
   * Hepatic metastases (unilateral or bilateral less than or equal to 5 lesions, less than or equal to 15 cm total diameter).
   * Primary peritoneal metastases (small disease load less than or equal to P2 disease) without massive ascites or intestinal obstruction.
   * Para-aortic lymph node metastases (stations 16 a1 and/or b2).
   * Lung metastases (less than or equal to 3 unilateral/bilateral, 9 cm total diameter).
   * Patients who present with both hepatic and peritoneal metastases must have no evidence of extensive para-aortic/retro-pancreatic lymph node metastases.
4. Greater than or equal to 18 years of age.
5. Must be able to understand and sign the Informed Consent Document.
6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) less than or equal to 2.
7. Life expectancy of greater than three months.
8. Patients of both genders must be willing to practice birth control during and for four months after receiving chemotherapy.
9. Hematology:

   * Absolute neutrophil count greater than 1300/mm^3 without the support of Filgrastim.
   * Platelet count greater than 75,000/mm^3.
   * Hemoglobin greater than 8.0 g/dl.
10. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 5 times the upper limit of normal. Except in the presence of obstructive liver metastases where ALT/AST may be up to 10 times the upper limit of normal.
    * Serum creatinine less than or equal to 1.5 mg/dl unless the measured creatinine clearance is greater than 60 mL/min/1.73 m^2.
    * Total bilirubin less than or equal to 2 mg/dl, except in the presence of obstructive metastases.
    * Prothrombin time (PT) within 2 seconds of the upper limit of normal (International Normalized Ratio (INR) less than or equal to 1.8).
11. No history of prior/other malignancies within the 2 years prior to enrollment with the exception of basal cell carcinoma.

EXCLUSION CRITERIA:

1. Prior treatment with 5-FU, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) (treatment with any of the components as separate regimens is allowable).
2. Inability to tolerate any of the chemotherapeutic agents.
3. Grade 2 or greater neuropathy.
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
5. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system; myocardial infarction; cardiac arrhythmias; obstructive or restrictive pulmonary disease.
6. Brain metastases or a history of brain metastases.
7. Childs B or C cirrhosis or with evidence of severe portal hypertension by history, endoscopy, or radiologic studies.
8. Weight less than 40 kg.
9. Significant ascites, greater than 1000cc in the absence of peritoneal disease.
10. History of congestive heart failure and/or an left ventricular ejection fraction (LVEF) less than 40%.

    Note: Patients at increased risk for coronary artery disease or cardiac dysfunction (e.g., greater than 65yo, diabetes, history of hypertension, elevated low-density lipoprotein (LDL), first degree relative with coronary artery disease) will undergo full cardiac evaluation and will not be eligible if they demonstrate significant irreversible ischemia on stress thallium or an ejection fraction < 40%.
11. Significant chronic obstructive pulmonary disease (COPD) or other chronic pulmonary restrictive disease with pulmonary function tests (PFT's) indicating an forced expiratory volume 1 (FEV1) less than 50% or a carbon monoxide diffusing capacity (DLCO) less than 40% predicted for age.

Note: Patients who have shortness of breath with minimal exertion or who are at risk for pulmonary disease (e.g., chronic smokers) will undergo pulmonary function testing and will not be eligible if their FEV1 is less than 50% of expected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07-22 (Actual); Primary Completion 2011-07-14 (Actual); Study Completion 2012-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Blazeby JM, Conroy T, Bottomley A, Vickery C, Arraras J, Sezer O, Moore J, Koller M, Turhal NS, Stuart R, Van Cutsem E, D'haese S, Coens C; European Organisation for Research and Treatment of Cancer Gastrointestinal and Quality of Life Groups. Clinical and psychometric validation of a questionnaire module, the EORTC QLQ-STO 22, to assess quality of life in patients with gastric cancer. Eur J Cancer. 2004 Oct;40(15):2260-8. doi: 10.1016/j.ejca.2004.05.023. PMID 15454251
- [Background] Sakamoto Y, Ohyama S, Yamamoto J, Yamada K, Seki M, Ohta K, Kokudo N, Yamaguchi T, Muto T, Makuuchi M. Surgical resection of liver metastases of gastric cancer: an analysis of a 17-year experience with 22 patients. Surgery. 2003 May;133(5):507-11. doi: 10.1067/msy.2003.147. PMID 12773978
- [Result] Rudloff U, Langan RC, Mullinax JE, Beane JD, Steinberg SM, Beresnev T, Webb CC, Walker M, Toomey MA, Schrump D, Pandalai P, Stojadinovic A, Avital I. Impact of maximal cytoreductive surgery plus regional heated intraperitoneal chemotherapy (HIPEC) on outcome of patients with peritoneal carcinomatosis of gastric origin: results of the GYMSSA trial. J Surg Oncol. 2014 Sep;110(3):275-84. doi: 10.1002/jso.23633. Epub 2014 Jul 5. PMID 25042700
- [Derived] Kemp CD, Kitano M, Kerkar S, Ripley RT, Marquardt JU, Schrump DS, Avital I. Pulmonary resection for metastatic gastric cancer. J Thorac Oncol. 2010 Nov;5(11):1796-805. doi: 10.1097/JTO.0b013e3181ed3514. PMID 20881648
- [Derived] Kerkar SP, Kemp CD, Duffy A, Kammula US, Schrump DS, Kwong KF, Quezado M, Goldspiel BR, Venkatesan A, Berger A, Walker M, Toomey MA, Steinberg SM, Giaccone G, Rosenberg SA, Avital I. The GYMSSA trial: a prospective randomized trial comparing gastrectomy, metastasectomy plus systemic therapy versus systemic therapy alone. Trials. 2009 Dec 23;10:121. doi: 10.1186/1745-6215-10-121. PMID 20030854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy | Systemic Chemotherapy Alone
Started | 8 | 7
Completed | 3 | 2
Not Completed | 5 | 5
Not completed — received some chemo, 4 and 9 cycles | 1 | 0
Not completed — not meet criteria for chemo foll surgery | 4 | 0
Not completed — progressed while on chemo | 0 | 2
Not completed — refused further treatment | 0 | 1
Not completed — withdrew consent | 0 | 1
Not completed — non-compliant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy | Systemic Chemotherapy Alone | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.73 (14.88) | 52.94 (11.67) | 49.33 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 3 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Patients With Limited Metastatic Gastric Carcinoma: Arm I
Description: Time between the first day of treatment and the date of death.
Time Frame: 12 weeks up to 3 years
Population: Patient #7 - alive 14 months at time of study closure; patient 11 alive 12 months at time of study closure; patient 15 expired following surgery.
Measure: Number; unit: Months
Groups:
- Surgery + HIPEC + Systemic Chemotherapy: Surgery -gastric resection, metastasectomy, and heated intraperitoneal chemotherapy (HIPEC) with Fluouracil (5-FU) 400 mg/m^2 intravenous (IV) over 5 minutes. Leucovorin 20 mg/m^2 IV and Oxaliplatin 460 mg/m^2 diluted in 2.0 L/m^2 of dextrose 5% in water (D5W) given as a heated intraperitoneal perfusion.
  Systemic chemotherapy - Irinotecan 165 mg/m^2 IV over 90 minutes, Oxaliplatin 85 mg/m^2 over 120 minutes, Leucovorin 200 mg/m^2 IV 120 minutes, 5FU 3200 mg/m^2 continuous IV infusion over 48 hours.
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy
Number analyzed (Participants) | 8
Months
  Patient #1 | 19
  Patient #2 | 11
  Patient #4 | 11
  Patient #6 | 4
  Patient #7 | 14
  Patient #9 | 5
  Patient #11 | 12
  Patient #15 | 0

2. Primary Outcome: Overall Survival in Patients With Limited Metastatic Gastric Carcinoma: Arm II
Description: Time between the first day of treatment and the date of death
Time Frame: 12 weeks up to 3 years
Population: Patient #3 - alive 17 months at time of study closure; patient 5 alive 6 months at time of study closure; patient 13 alive 8 months at time of study closure; patients 10,12 randomized but withdrew/no treatment; patient 14 randomized but did not return for treatment and lost to follow up. Patient #16 was lost to follow up after being randomized.
Measure: Number; unit: Months
Arm/Group | Systemic Chemotherapy Alone
Number analyzed (Participants) | 7
Months
  Patient #3 | 17
  Patient #5 | 6
  Patient #8 | 10
  Patient #10 | 0
  Patient #12 | 0
  Patient #13 | 8
  Patient #14 | 0

3. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 40.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy | Systemic Chemotherapy Alone
Number analyzed (Participants) | 8 | 7
Participants | 8 | 5

4. Secondary Outcome: 12 Months Disease Free Survival (DFS)
Description: Participants who were alive and disease free at 12 months. DFS was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response was disappearance of all target lesions. Partial response was at least a 30% decrease in target lesions. Progression was at least a 20% increase in target lesions and stable disease is neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy | Systemic Chemotherapy Alone
Number analyzed (Participants) | 8 | 7
Participants | 2 | 0

5. Secondary Outcome: Gillys Stage Before and After Surgery
Description: Gillys stage measures the completeness of the cytoreduction and is recorded before and after surgery. It is used to classify disease burden and determine prognosis. Stage 0 is no macroscopic signs of disease, stage 1 is nodules >5mm in one part of the abdomen, stage 2 is nodules >5 mm throughout the abdomen, stage 3 is nodules 5mm to 2 cm, and stage 4 is nodules < 2 cm.
Time Frame: Day 1
Measure: Number; unit: Stage
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy
Number analyzed (Participants) | 8
Stage
  Patient 1 Before Surgery | 0
  Patient 1 After Surgery | 0
  Patient 2 Before Surgery | 1
  Patient 2 After Surgery | 0
  Patient 3 Before Surgery | 0
  Patient 3 After Surgery | 0
  Patient 4 Before Surgery | 3
  Patient 4 After Surgery | 1
  Patient 5 Before Surgery | 0
  Patient 5 After Surgery | 0
  Patient 6 Before Surgery | 0
  Patient 6 After Surgery | 0
  Patient 7 Before Surgery | 1
  Patient 7 After Surgery | 0
  Patient 8 Before Surgery | 3
  Paitent 8 After Surgery | 0

6. Secondary Outcome: Completeness of Cytoreduction (CCR) Score
Description: CCR is assessed by Sugarbaker's criteria. CCR-0 is no residual tumor. CCR-1 is no residual nodules greater than 2.5 mm in diameter, CCR-2 is no residual nodules greater than 25 mm, and CCR-3 is residual nodules greater than 25 mm.
Time Frame: Day 1
Measure: Number; unit: Scores on a scale
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy
Number analyzed (Participants) | 8
Scores on a scale
  Patient 1 | 0
  Patient 2 | 0
  Patient 3 | 0
  Patient 4 | 2
  Patient 5 | 0
  Patient 6 | 0
  Patient 7 | 0
  Patient 8 | 0

7. Secondary Outcome: Median Blood Loss During Surgery
Description: Blood loss during surgery is related to complexity of the operation and via that to the stage of disease (more tumor to be cytoreduced, more blood loss).
Time Frame: Day 1
Measure: Median (Full Range); unit: ml
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy
Number analyzed (Participants) | 8
ml | 650 [400 to 2,800]

8. Secondary Outcome: Median Hospital Stay After Initial Surgery
Description: Recuperation period following complex surgery for this disease.
Time Frame: 1-10 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy
Number analyzed (Participants) | 8
Days | 17 [7 to 42]

9. Secondary Outcome: Median Duration of Cytoreduction Surgery and Heated Intraperitoneal Chemotherapy (HIPEC)
Description: Time it takes to perform this complex surgery and HIPEC to reduce tumor burden overall in this disease.
Time Frame: up to 12 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy
Number analyzed (Participants) | 8
hours | 10.1 [5 to 12]

10. Secondary Outcome: Quality of Life (QOL) Parameters Between the Two Study Groups
Description: QOL tools Functional Assessment of Cancer Therapy - Gastric cancer (FACT-Ga) specifically developed for the assessment of QOL in gastric cancer patients.
Time Frame: up to 3 years
Population: Zero participants were analyzed because data collected was insufficient due to the small sample size (I.e. too few patients to analyze) to make any comparisons that might be interpretable and subject to statistical rigor. Outcome will not be explored further.
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy | Systemic Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Patterns of Disease Recurrence Between the Two Therapeutic Approaches and Their Clinical Implications
Description: Compare surgery + heated intraperitoneal chemotherapy + systemic chemotherapy; and systemic chemotherapy alone to determine how each group responds clinically.
Time Frame: up to 3 years
Population: as for outcome 10
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy | Systemic Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 40.5 months.
Arm/Group | Surgery + HIPEC + Systemic Chemotherapy | Systemic Chemotherapy Alone
All-Cause Mortality (participants affected / at risk) | 7/8 | 7/7
Serious Adverse Events (participants affected / at risk) | 8/8 | 1/7
Other Adverse Events (participants affected / at risk) | 8/8 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery + HIPEC + Systemic Chemotherapy (N=8) | Systemic Chemotherapy Alone (N=7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Infections and infestations) | 2 (2) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >=38.5 degrees C)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Hemorrhage, GI:Peritoneal cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection: Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0x10e9/L):Blood
Infection: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0x10e9/L):Lung (pneumonia)
Infection: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0x10e9/L):Pelvis NOS
Infection with unknown ANC: Wound (Infections and infestations) | 1 (1) | 0 (0)
Leak (including anastomotic), GI: Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leak (including anastomotic), GI: Pancreas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Obstruction, GI:Small bowel NOS (Gastrointestinal disorders) | 2 (2) | 0 (0)
PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain:Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perforation, GI:Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 2 (2) | 0 (0)
Obstruction, GU:Ureter (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery + HIPEC + Systemic Chemotherapy (N=8) | Systemic Chemotherapy Alone (N=7)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Distention, bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Neurology - Other (Specify, tingling hands/feet) (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Pain:Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 1 (1)
Phosphate, serum-low (hypophospatemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (7) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (11)
Weight loss (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-05-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT00941655/Prot_SAP_000.pdf
  • Informed Consent Form (2012-05-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT00941655/ICF_001.pdf